CLINICAL TRIAL: NCT01498666
Title: Efficacy of Lactobacillus Reuteri Protectis on Functional Abdominal Pain (FAP) in Children 8-14 Years Old
Acronym: LactoFAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment rate was too slow according to study protocol and agreement.
Sponsor: BioGaia AB (Industry)
Collaborators: Sprim CRO, Italia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Q-PRE-0111-CLI-018
Record Dates: First submitted 2011-12-19; First posted 2011-12-23 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2013-12

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L. reuteri protectis tablets (Experimental): one tablet a day for 4 weeks
  Interventions: Dietary Supplement: L. reuteri protectis
- Placebo tablet (Placebo Comparator): one tablet a day for 4 weeks
  Interventions: Dietary Supplement: Placebo tablet

INTERVENTIONS:
Dietary Supplement: L. reuteri protectis — 1 tablet once daily for 4 weeks
  Arms: L. reuteri protectis tablets
Dietary Supplement: Placebo tablet — 1 tablet once daily for 4 weeks
  Other Names: Placebo
  Arms: Placebo tablet

SUMMARY:
The present clinical trial will examine the use of L. reuteri Protectis in children with functional abdominal pain. The aim of the study is to evaluate the use of L. reuteri Protectis on pain (severity and frequency) in children of 8-14 years old and with diagnosis of functional abdominal pain (FAP).

DETAILED DESCRIPTION:
Subject will be asked to consume a tablet every day for 4 weeks. Supplementation will be stopped after 4 weeks, and the subjects will be followed up for an additional 4 weeks. The subjects will complete a diary to record frequency and intensity of pain, use of medication, deviation from the usual diet, physical activities, and absence from school and other activities. Gastrointestinal symptoms are assessed.

ELIGIBILITY:
Inclusion Criteria:

* FAP (Functional Abdominal Pain) according to Rome III criteria for
* Child/Adolescent (Rasquin, 2006);
* 1 or more abdominal pain episodes per week over the past 8 weeks;
* Informed consent by study participant and at least one parent / legal guardian;
* Age 8-14 years;
* Pain severity at study entry must be at least 40 mm on a 100 mm VAS scale;
* Ability to understand and comply with the requirements of the trial;
* Stated availability throughout the study period.

Exclusion Criteria:

* Chronic illness;
* Surgery of Gastrointestinal tract;
* Any organic symptoms and/or clinical signs of disorder or disease other than FAP;
* Weight loss of 5% or more in body weight over the preceding 3 months;
* Any abnormal result of laboratory assays, also including screening for celiac disease, lactose intolerance;
* Exposure to any drug or medication (antidepressants, SSRIs, laxatives) in the past 3 months or regular use of this medication;
* Exposure to probiotics or antibiotics within 4 weeks prior to study; subjects can be included following a wash-out period of 4 weeks.
* Participation in other clinical trials in the past 3 months;
* Subjects with anemia;
* Subjects with special dietary needs

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint | 4 weeks
  Pain frequency measured by a subject diary, in the L. reuteri Protectis group and the placebo group, expressed as area under the pain-frequency curve and comparing L. reuteri Protectis vs. placebo over the 4-week supplementation period.

SECONDARY OUTCOMES:
Secondary endpoint | 56 days
  Pain frequency measured by subject diary and expressed as area under the curve, comparing L. reuteri protectis vs. placebo over the initial 2 weeks of the supplementation period. Pain severity measured by the face score system by Wong-Baker at day 14, 28 and 56 (follow up) vs baseline, and area under the curve for weeks 1-4 and 1-2. Treatment success, defined as ≥ 50% reduction in pain frequency in weeks 1-4. Reduction in days of absence from school. Parents' absence from work. Need of rescue medication.

CONTACTS AND LOCATIONS:
Overall Officials: Costantino DeGiacomo, MD, Principal Investigator — Niguarda Hospital
Locations (2):
- Italy (2):
  - AO Niguarda Ca' granda, Milan
  - AO "San Paolo", Milan